CLINICAL TRIAL: NCT07362394
Title: Autologous Dentine Graft Compared to Xenograft in Managing Periodontally Compromised Second Molar After Third Molar Removal - A Split-Mouth Randomized Controlled Trial
Brief Title: Autologous Dentine Graft Compared to Xenograft in Managing Periodontally Compromised Second Molar After Third Molar Removal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Nik Madihah Nik Aziz, Lecturer and Clinical Specialist in Periodontology, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UKM-FGG-ADG25; RSCH ID-25-08139-VWQ (Other: Malaysia National Medical Research Register)
Record Dates: First submitted 2025-12-27; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Impacted Mandibular Third Molar Extraction; Dentin Graft; Xenograft; Bone Defects
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a prospective, double-blinded, split-mouth, randomised controlled trial to evaluate the efficacy of autologous dentine grafts (ADGs) compared to commercially available xenografts in promoting periodontal and alveolar bone healing at distal surface of M2s following the surgical removal of impacted mandibular M3s.
  Participants will be enrolled in a randomised split-mouth design. In each patient, one extraction socket (control site) will be grafted with a commercially available xenograft material, while the contralateral socket (test site) will be grafted with an ADG, prepared intraoperatively from the patient's own extracted M3.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADG Group (Experimental): ADG will be immediately packed into the extraction socket against the distal root of M2 until cementoenamel junction (CEJ) level, before flap repositioning and suturing.
  Interventions: Biological: Autologous dentin graft
- Xenograft Group (Active Comparator): Xenograft will be placed using the same placement technique as that employed in the ADG group.
  Interventions: Biological: Xenograft

INTERVENTIONS:
Biological: Autologous dentin graft — Extracted mandibular M3 will be mechanically processed intraoperatively into dentine particles using the BonMaker® device (Korea Dental Solutions Co. Ltd., South Korea), in accordance with the manufacturer's instructions for chairside preparation of ADG.
  Other Names: Autogenous dentin graft; autogenous tooth bone graft; demineralised dentin matrix
  Arms: ADG Group
Biological: Xenograft — Commercially available xenograft, which is of bovine derivative
  Arms: Xenograft Group

SUMMARY:
The goal of this study is to evaluate the efficacy of autologous dentin graft (ADG) in treating periodontal defects on the distal aspect of mandibular 2nd molar (M2) after surgical removal of impacted mandibular 3rd molar (M3) by improving periodontal and radiological outcomes when compared with a xenograft, which is commercially available. The main questions it aims to answer are:

1. How does the clinical efficacy of ADG compare to xenografts, regarding wound healing and periodontal parameters at the distal aspect of periodontally compromised mandibular M2 following impacted M3 extraction?
2. How does the radiological bone regeneration at ADG-grafted sites differ from that at xenograft-grafted sites?
3. How do the post-operative patient-reported outcomes at sites receiving ADG differ from those at sites receiving xenografts?

Researchers will compare ADG to xenograft to see if ADG is more efficacious in managing periodontal defects on distal aspect of M2 after surgical removal of M3.

Participants will

1. Undergo bilateral surgical removal of M3 under general anaesthesia
2. Receive ADG on test site and xenograft on contralateral control site
3. Come back for clinical assessments, wound healing assessments and radiographic assessments for 5 times after the surgery (2 weeks, 1 month, 3 months, 6 months and 12 months)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 26 years and above who can give informed consent and are scheduled for bilateral surgical removal of mesioangular or horizontally impacted mandibular M3s
* Present with a periodontally compromised mandibular second molar, defined by the presence of probing pocket depth (PPD) greater than 4 mm on the distal aspect
* Type of impaction of M3s on both sides must be symmetrical
* Consent to the use of xenograft as control

Exclusion Criteria:

* Smokers
* Poor oral hygiene with >30% full mouth plaque score (FMPS)
* Pregnant or lactating mothers
* Have uncontrolled systemic conditions such as diabetes or immunodeficiency disorders
* On medications that affect bone metabolism, including bisphosphonates or corticosteroids
* History of periodontal surgery or grafting at the intended surgical site
* Presence of acute infection and M2s with distal caries and Grade III mobility

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Assessment | Baseline, 3 months, 6 months, 12 months
  Probing pocket depth (PPD) (mm)
Clinical Assessment | Baseline, 3 months, 6 months, 12 months
  Clinical attachment level (CAL) (mm)
Radiographic Assessment | Baseline, 6 months, 12 months
  Osseous defect depth (ODD)

SECONDARY OUTCOMES:
Wound Healing Assessment | Baseline, 2 weeks, 1 month, 3 months, 6 months and 12 months
  Landry Wound Healing Index
Patient Reported Outcome Measures | Baseline, Day 1, Day 3, 1 week, 2 weeks, 1 month
  Visual Analogue Scales (VAS) will be used to capture post-operative pain. 100 mm VAS ruler will be used, where the scale is from 0 (no pain) to 100 (worst pain imaginable).
Patient Reported Outcome Measures | Baseline, Day 1, Day 3, 1 week, 2 weeks, 1 month
  Pain Intensity Score from the Malay validated version of the Brief Pain Inventory (BPI) questionnaire will be used. This section consists of 4 questions where the scale is from 0 (no pain) to 10 (worst pain imaginable).
Patient Reported Outcome Measures | Baseline, Day 1, Day 3, 1 week, 2 weeks, 1 month
  Pain Interference Score from the Malay validated version of the Brief Pain Inventory (BPI) questionnaire will be used. This section consists of 7 questions where the scale is from 0 (does not interfere) to 10 (completely interferes).

OTHER OUTCOMES:
Clinical Assessment | Baseline, 1 month, 3 months, 6 months, 12 months
  Plaque index (PI)(%)
Clinical Assessment | Baseline, 1 month, 3 months, 6 months, 12 months
  Bleeding on probing (BOP)(%)
Radiographic Assessment | Baseline, 6 months, 12 months
  Advanced radiomic analysis will be conducted using LifeX, a dedicated and validated radiomics software platform, to extract detailed quantitative features of trabecular bone microarchitecture, expressed in the form of grayscale value.

CONTACTS AND LOCATIONS:
Locations (1):
- Kuala Lumpur Hospital, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
To protect confidentiality of study subjects